CLINICAL TRIAL: NCT02890550
Title: Clinical Study of a Single Ciliopathy: Alström Syndrome
Status: Terminated | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5514
Record Dates: First submitted 2016-08-19; First posted 2016-09-07 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Alström Syndrome (ALMS)
Keywords: Ciliopathy; Retinitis pigmentosa; ALMS1 gene
MeSH Terms: conditions — Alstrom Syndrome; Ciliopathies; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, urine, tissue (skin biopsy, adipose tissue)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 30 Patients Alström syndrome
- 60 Related patients Alström syndrome

SUMMARY:
The aim of the study is to characterize the clinical manifestations of ALMS within the ciliopathies to prevent complications and determine preventive and therapeutic targets.

The investigators believe that the clinical consequences of mutations in the gene result ALMS1 unprecedented protests and the ALMS study should help to be informed, not only about the understanding and decision support other ciliopathies, but also about some common diseases, as some physiopathogenic roads could be common; the rare disease being exacerbated a model of the channel concerned. Secondarily, the clinical data generated by this project will also be used as part of basic research (eg comparison with results in animal models, use of human cells for in vitro studies or transcriptomic ....) (which will be a secondary upgrading to this work).

ELIGIBILITY:
Inclusion Criteria for Patients with Alström syndrome:

* Age> 2 years
* Affiliated with a social security scheme
* Informed consent signed
* Retinal dystrophy and proved at least three diagnostic criteria Alström syndrome (Criteria Marshall et al, 2005):
* Early obesity
* Deafness
* Dilated cardiomyopathy
* Type 2 diabetes
* Hypogonadism
* Absence of polydactyly
* Lack of mental retardation
* A family history of the ALMS
* Mutation in the ALMS gene identified

Inclusion Criteria for Related of Alström patients :

* Father / Mother of a patient diagnosed with Alström
* Age greater than 18 years
* Affiliated with a social security scheme
* Informed consent signed

Exclusion Criteria for Patients with Alström syndrome:

* Current pregnancy (a pregnancy test is routinely performed at baseline)
* Pregnant or breastfeeding women
* Intercurrent diseases do not allow the practice exams in protocol
* Subject to exclusion period (determined by a previous study or a study in progress)

Exclusion Criteria for Related of Alström patients :

* Age less than 18 years
* Subject to exclusion period (determined by a previous study or a study in progress)

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited through the investigators' consultation Reference Center for Rare Diseases in Ophthalmological Genetics (CARGO) or sent by their colleagues from other cities including through very geneticists genetic Group or 3rd Thursdays ophthalmologists colleagues. Prior consultation CARGO will disclose the medical records of the intention of the patient to participate in this research (source document).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-04; Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Genetic Diagnosis | 6 months
  In this project, 8 clinical research modules covering major medical issues goshawks ALMS (Genetic diagnosis, neurosensory infringement (ophthalmology and ENT (hearing and olfaction) and neuro-cognitive impairment), obesity & diabetes, endocrine achievement, nephrologic achievement, cardiological achievement, pneumologic achievement, reproductive biology). For each module, the current state of knowledge, clinical issues and their impact on the management of short and medium term ALMS patients are detailed. The clinical complications of this disease must be identified rationally and treatment and clinical management optimized on robust foundations for enhanced medical knowledge. The development of targeted therapies will depend on the clinical research data is the basic foundation of work which can then be enriched by the scientific data currently booming in this area.
Neurosensory infringement | 6 months
  * Ophtalmology study: consultation with visual acuity evaluation, examination at the slit lamp, intraocular pressure measurement, fundus examination, evaluation of Goldmann visual field, rétinophotography, standard and multifocal electroretinography, color vision, Optical Coherence Tomography (OCT), orthoptic balance
    * proportion of initial macular involvement and impact on future therapeutic trials (eg retina / age thickness)
    * consequences of low vision on posterior optical channels (including occipital cortex)
  * Olfaction study: brushing the nasal mucosa, isotopic mucociliary clearance, olfactometry (test UPSIT) gustometry, audiogram, otoacoustic emissions, auditory evoked potentials
    * Is the origin of deafness endocochlear only?
    * OAS are they a predictive test and prognosis?
    * Are ALMS patients suffering anosmia as for other ciliopathies?
    * Mobile eyelashes respiratory mucosal abnormalities are they like other ciliopathies?
Neurocognitive impairment | 6 months
  Neurocognitive explorations:
  * Neuropsychological assessment with cognitive tests, psychiatric evaluation, MRI, to determine if ALMS patients have cognitive impairment.
  * Validation of a second population of a new innovative battery of neurocognitive tests for the visually impaired.
Obesity - Diabetes | 6 months
  Study of the origin of obesity:
  * Origin central or peripheral obesity?
  * Determinism of insulin resistance and diabetes? nutrition consultation, impedance, basal calorimetry and OGTT, food investigation over 3 days and dietary questionnaires, laboratory tests, calorimetry, polysomnography (Embletta), abdominal-pelvic MRI
Endocrine Achievement | 6 months
  Endocrine study:
  - Determine the primary endocrine deficiencies of those who are secondary to obesity and metabolic disorders.
  OGTT, test LHRH
Nephrologic achievement | 6 months
  Nephrology consultation including water deprivation test and renal ultrasound, to determine what is the primum movens at the renal impairment (glomerular or tubular origin), and if there is a particular component in fibrotic renal disease compared to other ciliopathies.
  nephrology consultation, water deprivation test, renal ultrasound
Cardiological achievement | 6 months
  Study of cardiovascular risk factors:
  - Which patients have cardiac fibrosis? At what age and what connection with possible cardiomyopathy childhood? Cardiology consultation including echocardiogram, electrocardiogram (ECG), ambulatory blood pressure measurement, cardiac MRI, cardiac great vessels holter doppler
Pneumologic achievement | 6 months
  Respiratory function study:
  * Are respiratory alterations related to a breach of mobile eyelashes?
  * Do ALMS patients develop respiratory fibrosis and in which context ? Spirometry, exhaled NO
Reproductive biology | 6 months
  To explain infertility of ALMS patients (men or women)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène DOLLFUS, MD, Principal Investigator — Centre de Référence pour les Affections Rares en Génétique Ophtalmologique (CARGO), Hôpitaux Universitaires de Strasbourg
Locations (14):
- France (14):
  - CMCO, Hôpitaux Universitaires, Schiltigheim
  - Centre d'Investigation Clinique, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Centre de Référence pour les Affections Rares en Génétique Ophtalmologique (CARGO), Hôpitaux Universitaires, Strasbourg
  - Clinique Psychiatrique, Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service de Cardiologie, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service de néphrologie et hémodialyse, Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service de physiologie et des Explorations Fonctionnelles, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service de Psychothérapie pour Enfants et Adolescents, Hôpital Civil, Hôpitaux Universitaires, Strasbourg
  - Service d'Imagerie 1, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg
  - Service d'ORL et de Chirurgie Cervico-Faciale, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg
  - Service de Génétique Médicale, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg
  - Service de Médecine Interne, Endocrinologie et Nutrition, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg
  - Service de Pédiatrie 1, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg
  - Service de Radiologie 2, Hôpital de Hautepierre, Hôpitaux Universitaires, Strasbourg

IPD SHARING:
Plan to Share IPD: No